CLINICAL TRIAL: NCT05142865
Title: A Phase II Clinical Study Evaluating the Safety and Efficacy of Camrelizumab Combined With Chemotherapy and Apatinib as First Line Treatment in Advanced or Metastatic Extrapulmonary Neuroendocrine Carcinomas（EP-NEC）
Brief Title: Camrelizumab Combined With Chemotherapy and Apatinib for Extrapulmonary Neuroendocrine Carcinomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, Professor, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-NEC-Ⅱ-001
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Advanced or Metastatic EP-NEC
MeSH Terms: interventions — camrelizumab; Etoposide; Carboplatin; Cisplatin; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+ Chemotherapy+Apatinib (Experimental): Induction stage：Camrelizumab 200 mg administered intravenously (IV) on Day 1 +Etoposide (100mg/m2 IV continuously on Day 1, 2 and 3）+Carboplatin（AUC 5 mg/mL/min IV on Day 1) or Cisplatin(25mg/m2，continuously on Day 1, 2 and 3) Q3W for 4-6 cycles; Maintenance stage：Camrelizumab 200 mg administered intravenously (IV) on Day 1 of each 21-day cycle plus Apatinib capsules 250 mg given orally, once daily in 21-day cycle .
  Interventions: Drug: Camrelizumab; Drug: Etoposide; Drug: Carboplatin; Drug: Cisplatin; Drug: Apatinib

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab intravenous infusion was administered at a dose of 200 mg on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4/6) and maintenance phase ,until PD.
  Other Names: SHR-1210
Drug: Etoposide — 100mg/m2 IV continuously on Day 1, 2 and 3 of each 21-day cycle during the induction phase (Cycles 1-4/6)
Drug: Carboplatin — AUC 5 mg/mL/min IV on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4/6)
Drug: Cisplatin — 25mg/m2，continuously on Day 1, 2 and 3 of each 21-day cycle during the induction phase (Cycles 1-4/6)
Drug: Apatinib — 250 mg given orally, once daily in 21-day cycle

SUMMARY:
This is an open-label，single-arm, phase II exploratory study that evaluates the efficacy and safety of Camrelizumab combined with Chemotherapy （carboplatin or cisplatin + etoposide）and Apatinib as First Line treatment in Advanced or Metastatic Extrapulmonary Neuroendocrine Carcinomas（EP-NEC）

ELIGIBILITY:
Inclusion Criteria:

- Eligible patients for this study must meet all of the following criteria:

1. Pathologically or cytologically diagnosed as locally advanced or metastases extrapulmonary neuroendocrine carcinoma that cannot be surgically removed.
2. Aged 18-75，male and female
3. Patients who have not received systemic treatment for advanced or metastatic EP-NEC . Subjects who have previously received adjuvant or neoadjuvant therapy (including chemotherapy, radiotherapy or radiochemotherapy) for EP-NEC must have completed the last dose at least 6 months before enrollment . Palliative radiotherapy is permitted, but it must be completed at least 2 weeks prior to the study treatment. The lesions in the irradiation field cannot be used as target lesions for efficacy evaluation, and radiotherapy-related adverse reactions must be restored to at least Grade 0-1.
4. ECOG PS 0-1.
5. At least 1 measurable lesion according to RECIST criteria.
6. Adequate organ and bone marrow function, defined as follows:

   * White blood cell count (WBC) ≥ 3,000/mm3 (3.0 × 109/L);
   * Absolute neutrophil count (ANC) ≥ 1,500/mm3 (1.5 × 109/L);
   * Platelet count (PLT) ≥ 100,000/mm3 (100 × 109/L);
   * Hemoglobin (Hb) ≥ 9 g/dL (90 g/L);
   * Serum albumin ≥ 3.0 g/dL (30 g/L);
   * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 ml/min;
   * Total bilirubin (BIL) ≤ 1.5 x ULN;
   * AST or ALT ≤ 2.5 x ULN, patients with liver metastases should ≤ 5×ULN; international normalized ratio (INR) ≤ 1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN;
   * Urine protein<2+; if the urine protein is ≥2+, the 24-hour urine protein must be ≤1g.
7. Subjects must agree and have signed the informed consent form, be willing and able to follow the scheduled visits, study treatment, laboratory tests, and other study procedures.
8. Life expectancy > 12 weeks.
9. Female subjects of childbearing age are not pregnant or breastfeeding and are strictly contraceptive.

Exclusion Criteria:

1. Presence of known uncontrolled or symptomatic active central nervous system (CNS) metastasis, manifested as clinical symptoms, cerebral edema, spinal cord compression, cancerous meningitis, leptomeningeal disease, and/or progressive growth. For CNS metastases that have been adequately treated, and neurological symptoms can return to baseline levels at least 2 weeks before enrollment (except for residual signs or symptoms related to CNS treatment), they can be included . In addition, subjects must stop corticosteroids or receive a stable dose of ≤ 10 mg/d or a gradually decreasing dose of prednisone (or an equivalent dose of other corticosteroids) at least 2 weeks before enrollment.
2. Have received the following treatments or drugs before enrollment:

   ① A major operation was performed within 28 days before enrollment (tissue biopsy and peripheral venipuncture for central venous catheterization [PICC]/infusion port implantation are allowed).

   ② Using immunosuppressive drugs within 7 days before enrollment, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroid hormones (no more than 10 mg/d prednisone or other corticosteroids with equivalent physiological doses)

   ③ within 28 days before enrollment or planned to receive live attenuated vaccine during the study period and 60 days after the end of study drug treatment.

   ④ Receive chemotherapy within 28 days before enrollment;
3. Prior malignancy within 3 years, except adequately treated basal cell carcinoma or squamous cell skin cancer ,superficial bladder cancer, cervical carcinoma in situ, breast ductal carcinoma in situ and papillary thyroid cancer.
4. Prescence of any active, known or suspected autoimmune diseases. Subjects who are in a stable state and do not require systemic immunosuppressive therapy are allowed, such as type I diabetes, hypothyroidism that only requires hormone replacement therapy, and skin diseases that do not require systemic therapy (eg, vitiligo, psoriasis disease and hair loss).
5. Prior treatment with anti-PD-1/PD-L1 antibodies, anti-PD-L2 antibodies, anti-CD137 antibodies, CTLA-4 antibodies, or other drugs/antibodies that act on T cell costimulation or checkpoint pathways.
6. Prescence of clinically significant bleeding symptoms or a clear bleeding tendency within 3 months before enrollment; gastrointestinal perforation and/or gastrointestinal fistula occurred within 6 months before enrollment; 6 before enrollment Arterial/venous thrombosis events that occurred within a month, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism.
7. Have major vascular disease (for example, an aortic aneurysm that requires surgical repair or recent peripheral arterial thrombosis) occurred within 6 months before the start of study treatment.
8. Severe, unhealed or dehisced wounds and active ulcers or untreated fractures.
9. Have intestinal obstruction and/or have clinical signs or symptoms of gastrointestinal obstruction within 6 months before the start of the study treatment.
10. Prescence of interstitial lung disease, non-infectious pneumonia or uncontrollable systemic disease.
11. Known to be allergic to the study drug or any of its excipients; or have a severe allergic reaction to other monoclonal antibodies.
12. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU/ml; hepatitis C,defined as HCV-RNA higher than the detection limit of the analytical method) or combined hepatitis B and C co-infection.
13. Any of the following conditions observed within 6 months prior to the enrollment: myocardial infarction, severe/unstable angina, NYHA grade 2 or higher cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmia, and symptomatic congestive heart failure exhaustion.
14. Hypertension, which cannot be well controlled by antihypertensive drugs (systolic blood pressure> 140 mmHg or diastolic blood pressure> 90 mmHg).
15. Systemic use of antibiotics for ≥ 7 days within 4 weeks before enrollment, or unexplained fever > 38.5 ° C during screening / before the first administration (according to the judgment of the investigator, fever caused by tumor can be enrolled) .
16. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
17. Participated in any other drug clinical research within 4 weeks before enrollment, or no more than 5 half-lives from the last drug use in the study. Known history of psychotropic drug abuse or drug abuse.
18. Subjects with other severe physical or psychiatric disorders or laboratory abnormalities, which may increase the risk of participating in this study or interfere with the study results, as well as those deemed unsuitable by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-14 (Estimated); Primary Completion 2024-01-14 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate （ORR） | 2 years
  Defined as percentage of participants achieving complete response (CR) and partial response (PR) assessed by the investigator according to the RECIST 1.1

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  OS is defined as the time from registration to death due to any cause.
Progression-Free Survival (PFS) | 3 years
  PFS is defined as the time from registration to the first documented disease progression or death due to any cause, whichever occurs first.
Duration of Response (DOR) | 3 years
  For participants who demonstrate CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters), DOR is defined as the time from first documented evidence of CR or PR until disease progression per RECIST 1.1 based on assessments by the investigator or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | 2 years
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or stable disease per RECIST 1.1
Adverse event (AE) | 2 years
  An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who experience an AE will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qiu, MD, Principal Investigator — Tongji Hospital; Yuhong Dai, MD, Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital，Tongji Medical College Affiliated，Huazhong University of Science ＆ Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No